CLINICAL TRIAL: NCT00446563
Title: An Open-label, Randomized, Parallel Group Study Comparing the Efficacy and Safety of Amlodipine in Combination With Valsartan Compared to Losartan in Combination With Hydrochlorothiazide Given for 52 Weeks on the Regression of Left Ventricular Hypertrophy in Patients With Mild to Moderate Hypertension
Brief Title: Efficacy and Safety of Valsartan in Combination With Amlodipine Compared to Losartan Plus Hydrochlorothiazide in Patients With Hypertension and Left Ventricular Hypertrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAA489ADE02
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension; Hypertrophy, Left Ventricular
Keywords: Left ventricular hypertrophy, hypertension, valsartan, amlodipine
MeSH Terms: conditions — Hypertension; Hypertrophy; Hypertrophy, Left Ventricular | interventions — Valsartan; Amlodipine; Hydrochlorothiazide; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amlodipine + Valsartan (Experimental): Participants received 160 mg Valsartan and 5 mg amlodipine orally once a day for 52 weeks. If blood pressure was not normalized at week 4, treatment was uptitrated to valsartan/amlodipine 160/10 mg. Participants with still uncontrolled hypertension could receive add-on antihypertensive medication.
  Interventions: Drug: Valsartan; Drug: Amlodipine
- Losartan + Hydrochlorothiazide (Active Comparator): Participants received 100 mg losartan and 12.5 mg Hydrochlorothiazide (HCT) orally once a day for 52 weeks. If blood pressure was not normalized at week 4, treatment was uptitrated to losartan/HCT 100/25 mg, respectively, until end of study. Participants with still uncontrolled hypertension could receive add-on antihypertensive medication.
  Interventions: Drug: Hydrochlorothiazide; Drug: Losartan

INTERVENTIONS:
Drug: Valsartan — 160 mg film coated tablets taken orally once daily in the morning.
  Arms: Amlodipine + Valsartan
Drug: Amlodipine — 5 mg or 10 mg tablets taken orally once daily in the morning.
  Arms: Amlodipine + Valsartan
Drug: Hydrochlorothiazide — 12.5 mg or 25 mg tablets taken orally once daily in the morning.
  Arms: Losartan + Hydrochlorothiazide
Drug: Losartan — 100 mg tablets taken orally once daily in the morning.
  Arms: Losartan + Hydrochlorothiazide

SUMMARY:
This study will evaluate the safety and efficacy of amlodipine plus valsartan in patients with hypertension and left ventricular hypertrophy

ELIGIBILITY:
Inclusion Criteria:

* Caucasian; male or female outpatients and age between 18-80 years of age, inclusive.
* Patients with a history of essential hypertension and who are actually treated either with an antihypertensive monotherapy and with a diastolic blood pressure >=90 and <= 105mmHg or with a combination therapy (limited to two active compounds) and with a diastolic blood pressure of >=90 and <= 100mmHg.
* Patients with Left Ventricular Hypertrophy

Exclusion Criteria:

* Severe hypertension
* Symptomatic heart failure
* History of stroke, heart attack, coronary bypass surgery etc.
* Insulin-dependent diabetes mellitus or poorly controlled diabetes mellitus.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- 25 centers in Germany, Ludwigshafen, Germany

REFERENCES:
- [Derived] Bruder O, Jensen CJ, Bell M, Rummel R, Boehm G, Klebs S, Sieder C, Senges J. Effects of the combinations of amlodipine/valsartan versus losartan/hydrochlorothiazide on left ventricular hypertrophy as determined with magnetic resonance imaging in patients with hypertension. J Drug Assess. 2011 Dec 16;1(1):1-10. doi: 10.3109/21556660.2011.639418. eCollection 2012. PMID 27536421

RESULTS

PARTICIPANT FLOW:
Groups:
- Valsartan and Amlodipine: Participants received 160 mg Valsartan and 5 mg amlodipine orally once a day for 52 weeks. If blood pressure was not normalized at week 4, treatment was uptitrated to valsartan/amlodipine 160/10 mg. Participants with still uncontrolled hypertension could receive add-on antihypertensive medication.
- Losartan and HCTZ: Participants received 100 mg losartan and 12.5 mg Hydrochlorothiazide (HCT) orally once a day for 52 weeks. If blood pressure was not normalized at week 4, treatment was uptitrated to losartan/HCT 100/25 mg, respectively, until end of study. Participants with still uncontrolled hypertension could receive add-on antihypertensive medication.
Period: Overall Study
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Started | 43 | 47
Completed | 36 | 38
Not Completed | 7 | 9
Not completed — Adverse Event | 4 | 3
Not completed — Abnormal laboratory value(s) | 0 | 1
Not completed — Abnormal test procedure result(s) | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Administrative problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ | Total
Number analyzed (Participants) | 43 | 47 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12.2) | 57.2 (10.9) | 57.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 31 | 34 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular Mass Index (LVMI) Measured Via Magnetic Resonance Imaging (MRI)
Time Frame: Baseline to week 52
Population: The intention-to-treat (ITT) population consisted of all patients who had a baseline MRI assessment. If patients dropped out prior to the scheduled observation period, every effort should have been taken to get a final MRI scan which could then be used for the ITT analysis.
Measure: Mean (Standard Deviation); unit: g/m˄2
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
g/m˄2 | -7.1 (16.50) | -9.1 (18.89)

2. Secondary Outcome: Change From Baseline to the End of Study in Left Ventricular Mass Index (LVMI) Normalized to Body Surface Area Assessed by MRI
Time Frame: Baseline to week 52
Population: The intention-to-treat (ITT) population consisted of all patients from the safety population who had a baseline MRI assessment. If patients dropped out prior to the scheduled observation period, every effort should have been taken to get a final MRI scan which could then be used for the ITT analysis.
Measure: Mean (Standard Deviation); unit: g/m˄2
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
g/m˄2 | -3.5 (7.4) | -4.4 (9.3)

3. Secondary Outcome: Change From Baseline to the End of Study in Interventricular Septum Thickness (IVS) Assessed by MRI
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
mm | -1.1 (1.5) | -0.6 (1.3)

4. Secondary Outcome: Change From Baseline to the End of Study in Posterior Wall Thickness Assessed by MRI
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
mm | -0.4 (1.1) | -0.3 (1.2)

5. Secondary Outcome: Change From Baseline to the End of Study in Left Ventricular Ejection Fraction (LVEF) Assessed by MRI
Description: Ejection fraction is a measurement of the percentage of blood that is pumped out of a filled ventricle with each heartbeat.
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
Percentage | -0.8 (6.7) | -0.4 (5.9)

6. Secondary Outcome: Change From Baseline to the End of Study in Left Ventricular End-diastolic Volume (LVEDV) Assessed by MRI
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
ml | 0.1 (19.9) | -6.4 (22.9)

7. Secondary Outcome: Change From Baseline to the End of Study in Left Ventricular End-diastolic Volume (LVEDV) Normalized to Body Surface Area Assessed by MRI
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
ml | 0.0 (9.6) | -3.0 (11.2)

8. Secondary Outcome: Change From Baseline to the End of Study in Left Ventricular End-Systolic Volume (LVESV) Assessed by MRI
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
ml | 0.4 (10.3) | -1.5 (10.3)

9. Secondary Outcome: Change From Baseline to the End of Study in Left Ventricular End-Systolic Volume (LVESV) Normalized to Body Surface Area Assessed by MRI
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
ml | 0.2 (5.1) | -0.8 (5.1)

10. Secondary Outcome: Change From Baseline to the End of Study in Left Atrial (LA) Area Assessed by MRI
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm˄2
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
cm˄2 | -0.6 (3.2) | -1.0 (4.5)

11. Secondary Outcome: Change From Baseline to the End of Study in the Ascending Aortic Diameter Assessed by MRI
Time Frame: Baseline to week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
mm | 0.1 (1.9) | -0.8 (1.6)

12. Secondary Outcome: Change From Baseline to End of Study in Levels of N-terminal Pro-B Type Natriuretic Peptide (NT-proBNP)
Time Frame: Baseline to week 52
Population: The safety population consisted of the sample of all randomized patients who applied study medication at least once.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
pg/ml | -4.5 (56.41) | -40.1 (74.09)

13. Secondary Outcome: Change From Baseline to End of Study in Levels of High-sensitivity C-reactive Protein (Hs-CRP)
Time Frame: Baseline to week 52
Population: The safety population consisted of the sample of all randomized patients who applied study medication at least once.
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
mg/l | 0.8 (6.09) | -2.1 (9.90)

14. Secondary Outcome: Percentage of Participants Achieving Target Blood Pressure at Week 52
Description: Target blood pressure defined as having a mean sitting systolic blood pressure (MSSBP) < 140 mm Hg and a mean sitting diastolic blood pressure (MSDBP) < 90 mm Hg.
Time Frame: Week 52
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
Percentage of participants | 53.5 | 14.9

15. Secondary Outcome: Percentage of Participants Who Experienced Adverse Events (AEs)
Description: An adverse event was the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after obtaining informed consent even if the event was not considered to be related to study drug. Medical conditions/diseases present before obtaining informed consent were only considered adverse events if they worsened after study start. Abnormal laboratory values or test results constituted adverse events only if they induced clinical signs or symptoms, required study drug discontinuation or required therapy.
Time Frame: Baseline to week 52
Population: The safety population consisted of the sample of all randomized patients who applied study medication at least once.
Measure: Number; unit: Percentage of participants
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Number analyzed (Participants) | 43 | 47
Percentage of participants | 69.8 | 68.1

ADVERSE EVENTS:
Arm/Group | Valsartan and Amlodipine | Losartan and HCTZ
Serious Adverse Events (participants affected / at risk) | 2/43 | 6/47
Other Adverse Events (participants affected / at risk) | 15/43 | 16/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan and Amlodipine (N=43) | Losartan and HCTZ (N=47)
BRADYCARDIA (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1
VESTIBULAR NEURONITIS (Infections and infestations) | 0 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
THALAMIC INFARCTION (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan and Amlodipine (N=43) | Losartan and HCTZ (N=47)
DIARRHOEA (Gastrointestinal disorders) | 1 | 4
NAUSEA (Gastrointestinal disorders) | 1 | 3
OEDEMA PERIPHERAL (General disorders) | 4 | 0
BRONCHITIS (Infections and infestations) | 3 | 0
NASOPHARYNGITIS (Infections and infestations) | 3 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 2
HEADACHE (Nervous system disorders) | 0 | 3
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.